CLINICAL TRIAL: NCT02847468
Title: Multimetabolic 18F-Fluorodeoxyglucose (FDG) and 18F-Fluorocholine (FCH) Positron Emission Tomography (PET) as an Early Predictive Factor of Overall Survival in Patients With Advanced Hepatocellular Carcinoma Treated With Sorafenib
Acronym: PREMETHEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PREMETHEP
Record Dates: First submitted 2016-07-19; First posted 2016-07-28 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: FDG PET, FCH PET
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG and FCH PET (Experimental): Patients will performed a TEP with 2 different radiotracer before treatment is started and 1 month after treatment has been started.
  Interventions: Other: FDG Positron Emission Tomography; Other: FCH Positron Emission Tomography

INTERVENTIONS:
Other: FDG Positron Emission Tomography — Subject will performed Positrons Emission tomography (PET) with 18F-Fluorocholine (FDG) before treatment with Sorafenib is started and 1 month after treatment started.
Other: FCH Positron Emission Tomography — Subject will performed Positrons Emission tomography (PET) with 18F-Fluorocholine (FCH) before treatment with Sorafenib is started and 1 month after treatment started.

SUMMARY:
Hepatocellular carcinoma (HCC) is the third cause of death by cancer. For patients with inoperable advanced HCC, systematic therapy with Sorafenib, a multikinase inhibitor that has both antiangiogenic and antiproliferative effect, is the only therapeutic with proven survival benefits. However, the efficacy of Sorafenib remains inconstant with a media overall survival of 10,7 months and a disease control rate only 35 to 43%; moreover, the overall incidence of treatment-related adverse event is 80%. Thus, it appears essential to find an early and accurate way to determine which patients are best responding to therapy in order to avoid the toxicity and cost of ineffective therapy.

Positron Emission Tomography (PET) with 18F-Fluorodeoxyglucose (FDG) has shown limited performance in the setting of HCC because of lack of sensitivity, in particular for well-differentiated tumours. However FDG uptake is related to proliferation rate and is an efficient marker survival following liver transplantation and selective internal radiation therapy. Moreover, the addition of a dynamic first-pass acquisition to the standard static scan provides better characterization of the tumour by adding information on tumour perfusion.

FCH which reflects lipids metabolism and specifically choline kinase activity, has shown promising results for detection of HCC when compared with FDG alone. Moreover, choline activity is related to a kinase pathway in mammalian cells, which is specifically inhibited by Sorafenib. However FCH uptake remains inconstant in HCC, and is related to tumour differentiation, by opposition to FDG. Therefore, several studies have suggested that combined evaluation of tumour glucose and lipid metabolism could play a complementary role for the evaluation of HCC in the setting of detection, staging and to predict recurrence following surgical resection. Thus, the investigator hypothesize that the combination of FDG and FCH may be the most accurate imaging evaluation of HCC.

Thus the aim of the present study is to determine the predictive performance of survival of lipid and glucose metabolism and perfusion changes during Sorafenib therapy in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Inoperable (advanced or metastatic) HCC histologically proven, or diagnosed according to the Barcelona criteria, determined to be candidate for Sorafenib therapy
* Lesion(s) able to be selected as targeted lesion(s) for modified RECIST criteria
* patient ineligible for curative treatment
* Child-Pugh liver function (platelet count superior or equal to 60X1 000 000 000per liter; haemoglobin superior or equal to 8,5g/dl
* Performance status more or equal to 2
* Able to lie still for 45min for PET/CT scanning
* Able to understand and willing to signa written informed consent document
* Affiliated to the French social security social or beneficiary to such a regimen

Exclusion Criteria:

* Uncontrolled intercurrent illness with short-term life-threatening
* Pregnant or nursing woman
* Patient candidate to local/curative therapy of HCC (surgery, radiofrequency, transarterial chemoembolization, other local therapy).
* History of myocardial infarction less than 6 months before inclusion, uncontrolled hypertension, symptomatic congestive heart failure, anti-arrhythmic therapy (other than beta-blockers or digoxine)
* History of digestive bleeding less than 30 days before inclusion
* history of liver transplantation
* Previous treatment including Sorafenib Uncontrolled diabetes History of allergic reactions attributed to compounds of similar chemical or biologic composition to Fluorocholine, 18F-Fluorodeoxyglucose or Sorafenib
* Psychiatric illness/social situations that would limit compliance with the study requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Vital status | One year after study inclusion
  vital status will be death or alive

SECONDARY OUTCOMES:
Disease control | 4 months
  Absence of radiologic progression according to modified RECIST criteria
Questionnaire of quality of life (EORTC QLQ-C30) | 1 year
  Questionnaire will be completed by subject at each clinical surveillance visit

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, Pr, Study Director — Centre Georges François Leclerc
Locations (1):
- Emilie REDERSTORFF, Dijon, France

IPD SHARING:
Plan to Share IPD: No